CLINICAL TRIAL: NCT06468202
Title: Comparative Effectiveness of Two Aspirin Doses for Prevention of Hypertensive Disorders of Pregnancy: ASPIRIN TRIAL
Brief Title: Effectiveness of Two Aspirin Doses for Prevention of Hypertensive Disorders of Pregnancy: ASPIRIN TRIAL
Acronym: ASPIRIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Northwestern University (Other); Preeclampsia Foundation (Other)
Responsible Party: Principal Investigator, Maged Costantine, MD, MBA, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00079100
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hypertensive Disorders of Pregnancy; Preeclampsia; Gestational Hypertension
Keywords: Hypertensive disorders of pregnancy; Aspirin treatment; Pregnancy; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: A randomized double-blind, multicenter, comparative effectiveness trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants, providers, investigators or outcome assessors will know to which of these groups participants are assigned. In case of an emergency, however, the study doctor can get this information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 81 mg Aspirin (Experimental): Treatment A consisting of 81mg of aspirin (1 pill of 81mg & 1 matching placebo) daily
  Interventions: Drug: Aspirin 81 mg
- 162 mg Aspirin (Experimental): Treatment B consisting of 162mg of aspirin (2 pills, each of 81mg) daily
  Interventions: Drug: Aspirin 162 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Participants will be assigned to 81mg Aspirin
  Arms: 81 mg Aspirin
Drug: Aspirin 162 mg — Participants will be assigned to 162mg Aspirin
  Arms: 162 mg Aspirin

SUMMARY:
The overall goal of this large, pragmatic, comparative effectiveness trial is to test the hypothesis that among at-risk individuals, 162 mg/day aspirin is superior to 81 mg/day in preventing Hypertensive disorders of pregnancy (HDP), and that there are multiple factors associated with adherence with aspirin therapy that will be important to identify to enable optimal implementation of study findings and population-level benefits.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP), such as preeclampsia (PE) and gestational hypertension (gHTN), occur in ~15% of pregnant individuals, disproportionately affect self-identified non-Hispanic Black individuals (with the understanding that race is a socially defined construct and the inequity is related to social determinants of health), are increasing in frequency, and are associated with short- and long-term maternal and neonatal morbidities and mortality. There are currently no available therapeutics to treat individuals with HDP; thus, developing interventions for the prevention of HDP is of substantial public health significance. The U.S. Preventive Services Task Force (USPSTF) and other professional societies recommend or endorse the use of aspirin for prevention of HDP in individuals at high or moderate risk. However, there is great uncertainty regarding optimal dosing, whether there is heterogeneity of effectiveness of aspirin in reducing the risk of HDP among different populations, and what factors are associated with adherence.

The overall goal of this large, pragmatic, comparative effectiveness trial is to test the hypothesis that among at-risk individuals, 162 mg/day aspirin is superior to 81 mg/day in preventing HDP, and that there are multiple factors associated with adherence with aspirin therapy that will be important to identify to enable optimal implementation of study findings and population-level benefits. The trial will achieve the following specific aims:

Specific Aim 1: To compare the frequency of HDP (primary outcome), as well as other important secondary outcomes (gHTN, PE, preterm PE, PE-related adverse outcomes, aspirin-related safety outcomes, and patient-reported outcomes related to maternal health, pregnancy, and childbirth experiences) between the two aspirin treatment arms.

Specific Aim 2: To compare the gestational age at birth and the frequency of adverse perinatal outcomes (preterm birth, perinatal death, small-for-gestational-age birth, neonatal intensive care unit admission, and complications of prematurity), as well as patient-reported outcomes related to maternal-infant bonding between the two aspirin treatment arms.

Specific Aim 3: To use quantitative and qualitative analyses to elucidate facilitators and barriers associated with adherence to aspirin therapy in at-risk individuals during pregnancy in order to facilitate future implementation.

ELIGIBILITY:
Inclusion Criteria:

1. live intrauterine gestation ≤16 6/7 weeks gestational age based on best clinical obstetric estimate,
2. age 14 years or older and able to provide informed consent,
3. at least one of the following high-risk criteria: i) any prior pregnancy complicated by preeclampsia ii) current pregnancy complicated by chronic hypertension diagnosed before randomization (ACOG) iii) pre-gestational diabetes (on medication for diabetes prior to pregnancy, or diabetes is diagnosed prior to randomization with hemoglobin A1C of 6.5% or greater or abnormal 3-hour glucose tolerance test) iv) twin gestation (including higher order pregnancy reduced to twins prior to 14 weeks) v) chronic kidney disease vi) autoimmune disease (e.g., antiphospholipid syndrome, systemic lupus erythematous)
4. or two or more moderate-risk criteria for HDP (per USPSTF), i) nulliparity (no prior delivery at or after 20 weeks 0 days of gestation) ii) obesity (body mass index ≥30 kg/m2 at time of randomization) iii) age ≥35 years (at time of expected estimated due date) iv) Black race v) low income vi) personal risk factors (previous pregnancy with low birth weight or SGA infant, previous adverse pregnancy outcome [unexplained stillbirth], placental abruption, interval >10 years between pregnancies) vii) Family history of preeclampsia (i.e., mother or sister) viii) In vitro fertilization
5. patient not currently on aspirin OR patient on aspirin for obstetrical indications (e.g., related to IVF, or HDP) and: i- randomized before 130/7 weeks gestation, or ii- randomized on or after 13 0/7 weeks gestation and started aspirin within 2 weeks prior to randomization (e.g., aspirin started for HDP prevention at 12 0/7 weeks and patient randomized at 13 2/7 weeks).

Exclusion Criteria:

1. known allergy or hypersensitivity to aspirin or any medical condition where aspirin is contraindicated (e.g., active peptic ulcer disease, nasal polyps, NSAID-induced asthma, active gastrointestinal bleeding, known G6PD deficiency, severe hepatic dysfunction, bleeding disorders, history of bariatric surgery),
2. current or planned aspirin use in pregnancy for non-obstetrical indication (e.g., prior stroke/prior myocardial infraction),
3. age < 14 years,
4. involuntarily confined or detained,
5. considered as having a diminished decision-making capacity,
6. obstetrical ultrasound suspicious for major congenital abnormality, known or suspected fetal aneuploidy, fetal demise, or planned pregnancy termination,
7. participation in another trial that affects the primary outcome, without prior approval of the PI,
8. plan to deliver at an outside participating site with inability to obtain medical records,
9. monoamniotic twin gestation because of the risk of fetal demise and preterm delivery,
10. participation in this trial in prior pregnancy,
11. triplet or higher order pregnancy.

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 10742 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Hypertensive Disorder of Pregnancy (HDP) | From >20 weeks gestation until hospital discharge following delivery, up to 22 weeks
  HDP defined as preeclampsia or antepartum gHTN based on ACOG criteria

SECONDARY OUTCOMES:
Preeclampsia | From >20 weeks gestation until hospital discharge following delivery, up to 22 weeks
  preeclampsia based on ACOG criteria
Preterm preeclampsia | From >20 weeks and ≤ 36 weeks 6 days, up to 17 weeks
  Preeclampsia per ACOG criteria with delivery < 37 weeks'
Postpartum preeclampsia | From delivery weeks till 6 weeks postpartum; 6 weeks
  Postpartum preeclampsia per ACOG criteria
Gestational hypertension | From >20 weeks until onset of labor, up to 22 weeks
  Gestational hypertension per ACOG criteria
Severe maternal morbidity | From randomization up to 6 weeks postpartum, up to 48 weeks
  Need for intensive care, maternal admission to a hospital within the first 42 days postpartum for obstetric complications, or blood product transfusion
Core preeclampsia outcomes | From randomization up to 6 weeks postpartum, up to 48 weeks
  Composite and individual maternal outcomes (Mortality, Eclampsia, Stroke, Cortical blindness, Retinal detachment, Pulmonary edema, Acute kidney injury, Liver capsule hematoma, Placental abruption, Postpartum hemorrhage, Elevated liver enzymes, Thrombocytopenia, ICU admission, Mechanical ventilation)
Bleeding complications (maternal) | From randomization till delivery up to 36 weeks, up to 36 weeks
  Antepartum bleeding and Placental abruption
Bleeding complications (maternal) | From delivery till hospital discharge, up to 1 week
  Postpartum hemorrhage
Adherence to aspirin | From randomization until last day of medication intake, up to 42 weeks
  pill count
Preterm birth | At time of delivery
  Delivery <37 weeks
Gestational age at birth | At time of delivery
  Gestational age in weeks at time of delivery
Core offspring/neonatal outcomes | up to 6 weeks post-delivery
  Composite and individual neonatal outcomes (Stillbirth, SGA, Neonatal mortality, Neonatal seizures, Admission to NICU, Respiratory support)
Rate of SGA | At time of birth
  Rate of birthweight <10th percentile
Bleeding complications (neonatal) | Up to 6 weeks post-delivery
  Any neonatal intraventricular or intracranial hemorrhage
Complications of prematurity and neonatal safety outcomes | Up to 6 weeks post-delivery
  Composite of RDS, Grade III-IV IVH, PVL, Stage 2/3 NEC, BPD, Stage III or higher ROP, or early onset sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Maged Costantine, MD, MBA, Principal Investigator — Ohio State University; Denise Sholtens, PhD, Principal Investigator — Northwestern University Data Analysis and Coordinating Center
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - University of Mississippi, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio
  - University of Pittsburg Magee, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas, Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova HealthSystem, Falls Church, Virginia
  - Eastern Virginia Medical School - Old Dominion University, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No